CLINICAL TRIAL: NCT03259334
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Study of SHP647 as Induction Therapy in Subjects With Moderate to Severe Ulcerative Colitis (FIGARO UC 301)
Brief Title: Efficacy and Safety Study of SHP647 as Induction Therapy in Participants With Moderate to Severe Ulcerative Colitis
Acronym: FIGARO UC 301
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to discontinue the SHP647 (ontamalimab) clinical trial development program for inflammatory bowel diseases (IBD) early.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP647-301; 2017-000599-27 (EudraCT Number)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ontamalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ontamalimab 25 mg (Experimental): Participants will receive 25 milligrams (mg) of ontamalimab (SHP647) subcutaneous (SC) injection using a prefilled syringe (PFS) on Week 0, Week 4 and Week 8.
  Interventions: Drug: Ontamalimab
- Ontamalimab 75 mg (Experimental): Participants will receive 75 mg of ontamalimab (SHP647) SC injection using PFS on Week 0, Week 4 and Week 8.
  Interventions: Drug: Ontamalimab
- Placebo (Placebo Comparator): Participants will receive placebo matched to ontamalimab (SHP647) SC injection using PFS on Week 0, Week 4 and Week 8.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ontamalimab — Participants will receive 1 mL of SHP647 sterile aqueous buffered solution at an appropriate concentration to provide the intended dose of drug (25 or 75 mg).
  Other Names: PF-00547659; SHP647
  Arms: Ontamalimab 25 mg; Ontamalimab 75 mg
Other: Placebo — Participants will receive 1 mL of sterile aqueous buffered solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of SHP647 in inducing remission, based on composite score of participant-reported symptoms and centrally read endoscopy, in participants with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or their parent or legally authorized representative must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Participants must be able to voluntarily provide written, signed, and dated informed consent and/or assent, as applicable, to participate in the study.
* Participants must be between greater than or equal to (>=)16 and <=80 years of age at the time of the signing of the informed consent/assent form.
* Participants less than (<) 18 years of age must weigh >=40 kg and must have body mass index (BMI) >=16.5 kilogram per square meter (kg/m^2).
* Participants must have a documented diagnosis of UC for >=3 months before screening. The following must be available in each participant's source documentation:

  1. A biopsy report to confirm the histological diagnosis.
  2. A report documenting disease duration based upon prior colonoscopy. Note: If this documentation is not available at the time of screening, a colonoscopy with biopsy to confirm the diagnosis is required during the screening period.
* Participants must be willing to undergo a flexible sigmoidoscopy or colonoscopy, including biopsy sample collection, during screening after all other inclusion criteria have been met.
* Participants must have moderate to severe active UC, defined as a total Mayo score of >=6, including a centrally read endoscopic subscore >=2, rectal bleeding subscore >=1, and stool frequency subscore >=1 at baseline.
* Participants must have evidence of UC extending proximal to the rectum (ie, not limited to proctitis).
* Participants must have had an inadequate response to, or lost response to, or had an intolerance to at least 1 conventional treatment such as mesalamine (5-aminosalicylate [ASA]), glucocorticoids, immunosuppressants (azathioprine [AZA], 6-mercaptopurine [6-MP], or methotrexate [MTX]), or anti-tumor necrosis factor (TNF).
* Participants receiving any treatment(s) for UC are eligible provided they have been, and are anticipated to be, on a stable dose for the designated period of time.
* Participants are males or nonpregnant, nonlactating females who, if sexually active, agree to comply with the contraceptive requirements of the protocol, or females of nonchildbearing potential.

Exclusion Criteria:

- Participants with indeterminate colitis, microscopic colitis, non-steroidal anti-inflammatory drug-induced colitis, ischemic colitis, infectious colitis, or clinical/histologic findings suggestive of Crohn's disease.

* Participants with colonic dysplasia or neoplasia. (Participants with prior history of adenomatous polyps will be eligible if the polyps have been completely removed.)
* Participants with past medical history or presence of toxic megacolon.
* Participants with colonic stricture, past medical history of colonic resection, a history of bowel surgery within 6 months before screening, or who are likely to require surgery for UC during the treatment period.
* Participants at risk for colorectal cancer must have a colonoscopy performed during the screening period with results available within 10 days before the baseline visit, unless the participant has had a surveillance colonoscopy performed within 1 year prior to screening, and any adenomatous polyps found at that examination have been excised. Colonoscopy report and pathology report (if biopsies are obtained) from the colonoscopy performed during screening or in the prior year confirming no evidence of dysplasia and colon cancer must be available in the source documents.

Participants at risk for colorectal cancer include, but are not limited to:

1. Participants with extensive colitis for >=8 years or disease limited to left side of colon (ie, distal to splenic flexure) for >=10 years before screening, regardless of age.
2. Participants >=50 years of age at the time of signing of the informed consent form.

   - Participants have had prior treatment with SHP647.

   - Participants with known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients.

   - Participants have received anti-TNF treatment within 60 days before baseline.

   - Participants have received any biologic with immunomodulatory properties (other than anti-TNFs) within 90 days before baseline.

   - Participants have received any nonbiologic treatment with immunomodulatory properties (other than their current background UC treatment) within 30 days before baseline.

   - Participants have ever received anti-integrin/adhesion molecule treatment (example (eg): natalizumab, vedolizumab, efalizumab, etrolizumab, or any other investigational anti-integrin/adhesion molecule).

   - Participants have received parenteral or rectal glucocorticoids, or rectal 5-ASA, within 14 days before screening endoscopic procedure.

   - Participants have received leukocyte apheresis or selective lymphocyte, monocyte, or granulocyte apheresis or plasma exchange within 30 days before baseline.

   - Participants have participated in other investigational studies within either 30 days or 5 half-lives of investigational product used in the study (whichever is longer) before baseline.

   - Participants have received a live (attenuated) vaccine within 30 days before the baseline visit.

   - Participants with active enteric infections (positive stool culture and sensitivity), Clostridium difficile infection or pseudomembranous colitis [Participants with C. difficile infection at screening may be allowed re-test after treatment], evidence of active cytomegalovirus infection or Listeria monocytogenes, known active invasive fungal infections such as histoplasmosis or parasitic infections, clinically significant underlying disease that could predispose the participants to infections, or a history of serious infection (requiring parenteral antibiotic and/or hospitalization) within 4 weeks before the baseline visit.

   - Participants with abnormal chest x-ray findings at screening, such as presence of active tuberculosis, general infections, heart failure, or malignancy.

   - Participants with evidence of active or latent infection with Mycobacterium tuberculosis (TB) or participants with this history who have not completed a generally accepted full course of treatment before randomization are excluded. All other participants must have either the Mantoux (purified protein derivative [PPD]) tuberculin skin test or interferon gamma release assay (IGRA) performed.

Participants who have no history of previously diagnosed active or latent tuberculosis are excluded if they have a positive Mantoux (PPD) tuberculin skin test (ie >=5 millimeter [mm] induration) or a positive IGRA (the latter to be tested at the site's local laboratory) during screening or within 12 weeks before screening. If IGRA test cannot be performed locally, a central laboratory may be used, with prior agreement from the sponsor.

1. An IGRA is strongly recommended for participants with a prior Bacillus Calmette-Guerin (BCG) vaccination, but may be used for any participant. Documentation of IGRA product used and the test result must be in the participant's source documentation if performed locally. Acceptable IGRA products include QuantiFERON TB Gold Plus In-Tube Test.
2. If the results of the IGRA are indeterminate, the test may be repeated, and if a negative result is obtained, enrollment may proceed. In participants with no history of treated active or latent tuberculosis, a positive test on repeat will exclude the participant. Participants with a history of active or latent TB infection must follow instructions for "participants with a prior diagnosis of active or latent TB are excluded unless both of the following criteria are met" in this criterion.
3. Participants with repeat indeterminate IGRA results, with no prior TB history, may be enrolled after consultation with a pulmonary or infectious disease specialist who determines low risk of infection (ie, participant would be acceptable for immunosuppressant [eg, anti-TNF] treatment without additional action). This consultation must be included in source documentation.

Results from a chest x-ray, taken within the 12 weeks before or during screening must show no abnormalities suggestive of active TB infection as determined by a qualified medical specialist.

Participants with a prior diagnosis of active or latent TB are excluded unless both of the following criteria are met:

1. The participant has previously received an adequate course of treatment for either latent (eg, 9 months of isoniazid or an acceptable alternative regimen, in a locale where rates of primary multidrug TB resistance are <5%. Participants from regions with higher rates of primary multidrug TB resistance are excluded) or active (acceptable multidrug regimen) TB infection. Evidence of diagnosis and treatment must be included in source documentation. Consultation with a pulmonary or infectious disease specialist to confirm adequate treatment (ie, participant would be acceptable for immunosuppressant [eg, anti-TNF] treatment without additional action) must be performed during the screening period. The consultation report must be included in source documentation prior to enrollment.
2. A chest x-ray performed within 12 weeks before or during screening indicates no evidence of active or recurrent disease, and documentation of interpretation by a qualified medical specialist must be included in source documentation.

   * Participants with a pre-existing demyelinating disorder such as multiple sclerosis or new onset seizures, unexplained sensory motor, or cognitive behavioral, neurological deficits, or significant abnormalities noted during screening.
   * Participants with any unexplained symptoms suggestive of progressive multifocal leukoencephalopathy (PML) based on the targeted neurological assessment during the screening period.
   * Participants with a transplanted organ. Skin grafts to treat pyoderma gangrenosum are allowed.
   * Participants with a significant concurrent medical condition at the time of screening or baseline, including, but not limited to, the following:

<!-- -->

1. Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal (except disease under study), endocrine, cardiovascular, pulmonary, immunologic [eg, Felty's syndrome], or local active infection/infectious illness) that, in the investigator's judgment will substantially increase the risk to the participant if he or she participates in the study.
2. Cancer or history of cancer or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
3. Presence of acute coronary syndrome (eg, acute myocardial infarction, unstable angina pectoris) within 24 weeks before screening.
4. History of significant cerebrovascular disease within 24 weeks before screening.

   * Participants who have had significant trauma or major surgery within 4 weeks before the screening visit, or with any major elective surgery scheduled to occur during the study.
   * Participants with evidence of cirrhosis with or without decompensation.
   * Participants with primary sclerosing cholangitis.
   * Participants with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb).

Note: If a participant tests negative for HBsAg, but positive for hepatitis B virus (HBcAb), the participant would be considered eligible if no presence of HBV DNA is confirmed by HBV DNA polymerasechainreaction(PCR) reflex testing performed in the central laboratory.

- Participants with chronic hepatitis C (HCV) (positive HCVAb and HCVRNA). Note: Participants who are HCVAb positive without evidence of HCVRNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks prior to baseline]).

- Participants with any of the following abnormalities in hematology and/or serum chemistry profiles during screening.

Note: Screening laboratory tests, if the results are considered by the investigator to be transient and inconsistent with the participant's clinical condition, may be repeated once during the screening period for confirmation. Results must be reviewed for eligibility prior to the screening endoscopy procedure.

1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels >=3.0×upper limit of normal (ULN).
2. Total bilirubin level >=1.5×ULN or >2.0×ULN if the participant has a known documented history of Gilbert's syndrome.
3. Hemoglobin level <=80 gram per liter (g/L) (8.0 gram per deciliter [g/dL]).
4. Platelet count <=100×10^9 per liter (/L) (100,000 cells per cubic millimeter [mm^3]) or >=1000×10^9/L (1,000,000 cells/mm^3).
5. White blood cell count <=3.5×10^9/L (3500 cells/mm^3). - Absolute neutrophil count (ANC)<2×10^9/L (2000 cells/mm^3).

   * Serum creatinine level >1.5 × ULN or estimated glomerular filtration rate <30 ml/min/1.73m^2 based on the abbreviated Modification of Diet in Renal Disease Study Equation.

Note: If platelet count is <150,000 cells/mm^3, a further evaluation should be performed to rule out cirrhosis, unless another etiology has already been identified.

- Participants with known human immunodeficiency virus (HIV) infection based on documented history, with positive serological test, or positive HIV serologic test at screening, tested at the site's local laboratory in accordance with country requirements or tested at the central laboratory.

Note: A documented negative HIV test within 6 months of screening is acceptable and does not need to be repeated.

- Participants who have, or who have a history of (within 2 years before screening), serious psychiatric disease, alcohol dependency, or substance/drug abuse or dependency of any kind, including abuse of medical marijuana (cannabis).

- Participants with any other severe acute or chronic medical or psychiatric condition or laboratory or electrocardiogram (ECG) abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

* Female participants who are planning to become pregnant during study period.
* Participants who do not agree to postpone donation of any organ or tissue, including male participants who are planning to bank or donate sperm and female participants who are planning to harvest or donate eggs, for the duration of the study and through 16 weeks after last dose of investigational product.
* Participants who are investigational site staff members or relatives of those site staff members or Participants who are Shire employees directly involved in the conduct of study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (205):
- United States (37):
  - Atria Clinical Research - Clinedge - PPDS, Little Rock, Arkansas
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - Inland Empire Liver Foundation, Rialto, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Asthma and Allergy Associates PC - CRN - PPDS, Colorado Springs, Colorado
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Omega Research Consultants LLC - Clinedge - PPDS, Orlando, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - Gastrointestinal Diseases, Inc. Research, Columbus, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Medisphere Medical Research Center LLC, Evansville, Indiana
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - Clinical Trials of SWLA LLC, Lake Charles, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - New York Total Medical Care PC, Brooklyn, New York
  - Piedmont Healthcare, Statesville, North Carolina
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Consultants For Clinical Research Inc, Fairfield, Ohio
  - Allegheny Center For Digestive Health, Pittsburgh, Pennsylvania
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology-Union City, Union City, Tennessee
  - Inquest Clinical Research/Coastal Gastroenterology Associates, PA, Baytown, Texas
  - Northside Gastroenterology, Cypress, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - HP Clinical Research, Bountiful, Utah
  - Digestive Health Center at UWMC, Seattle, Washington
  - University of Washington, Seattle, Washington
  - CHI Franciscan Digestive Care Associates, Tacoma, Washington
  - Exemplar Research, Inc. - Elkins, Elkins, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Australia (7):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (7):
  - A.ö. Krankenhaus der Barmherzigen Brüder, Sankt Veit an der Glan, Carinthia
  - LKH-Universitätsklinikum Klinikum Graz, Graz, Styria
  - Klinikum Klagenfurt Am Woerthersee, Klagenfurt
  - Salzburger Landeskliniken, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Brazil (3):
  - Instituto Goiano de Gastroenterologia E Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, Santo André, São Paulo
- Croatia (8):
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - Opca Bolnica Karlovac, Karlovac, Karlovacka Županija
  - Opca bolnica Bjelovar, Bjelovar
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital Centre Split, Split
  - General Hospital Virovitica, Virovitica
  - General County Hospital Vukovar and Croatian Veterans Hospital, Vukovar
  - General Hospital Zadar, Zadar
- Czechia (6):
  - Hepato-Gastroenterologie HK, s. r. o., Hradec Králové, Královéhradecký kraj
  - PreventaMed s.r.o., Olomouc, Olomoucký kraj
  - Institut Klinicke A Experimentalni Mediciny, Prague
  - ISCARE I.V.F. a.s., Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
  - Nemocnice Pardubickeho kraje, a.s. Orlickoustecka nemocnice, Ústí nad Orlicí
- Germany (12):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Gastro Campus Research GbR, Münster, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Gastroenterologische Facharztpraxis am Mexikoplatz, Berlin-Zehlendorf
  - Sana Klinikum Biberach, Biberach an der Riss
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Westklinikum Hamburg Ggmbh, Hamburg
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, Munich
- Israel (6):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem
  - Galilee Medical Center, Nahariya
  - Nazareth EMMS Hospital, Nazareth
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
  - Baruch Padeh Poriya Medical Center, Tiberias
- Italy (15):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo (FG), Apulia
  - Azienda Ospedaliera Mater Domini Di Catanzaro, Catanzaro, Calabria
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
  - Azienda Ospedale Università Padova - Dipartimento Salute della Donna e del Bambino - INCIPIT - PIN, Padua, Veneto
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
  - A.O.U. Maggiore della Carità, Novara
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - La Sapienza-Università di Roma-Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Japan (17):
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaidô
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Jikei University Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Ome Municipal General Hospital, Ōme, Tokyo
  - Tokatsu Tsujinaka Hospital, Abiko-shi, Chiba
  - Hakodate Koseiin Hakodate Goryoukaku Hospital, Hakodate
  - Yuai Memorial Hospital, Koga
  - Kawabe Clinic, Koganei
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Hidaka Coloproctology Clinic, Kurume-shi
  - Aichi Medical University Hospital, Nagakute
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Onomichi General Hospital, Onomichi
  - Shiga University of Medical Science Hospital, Ōtsu
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Shinbeppu Hospital, Beppu, Ôita
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - Vilnius City Clinical Hospital, Vilnius
- Netherlands (5):
  - ETZ-Elisabeth, Tilburg, North Brabant
  - NWZ, location Alkmaar, Alkmaar, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - VU Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum Amsterdam, Amsterdam
- Poland (35):
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp.j.Specjalistyczne Centrum Gastrologii i Endoskopii Specj, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o., Włocławek, Kuyavian-Pomeranian Voivodeship
  - Krakowskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Lexmedica, Wroclaw, Lower Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lódz, Lódzkie
  - SPZOZ Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej UM w Lodzi, Lódz, Lódzkie
  - Instytut Centrum Zdrowia Matki Polki, Lódz, Lódzkie
  - Centrum Medyczne Warszawa - PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej VIVAMED, Warsaw, Masovian Voivodeship
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - H-T. Centrum Medyczne Endoterapia, Tychy, Silesian Voivodeship
  - Twoja Przychodnia - Szczecińskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Czestochowa - PRATIA - PPDS, Częstochowa
  - Centrum Medyczne Gdynia - PRATIA - PPDS, Gdynia
  - BioVirtus Centrum Medyczne, Józefów
  - Szpital Zakonu Bonifratrow pw. Aniolow Strozow w Katowicach, Katowice
  - NZOZ All Medicus, Katowice
  - Centrum Medyczne A-Z Clinic Mateusz Sidor, Piotr Puc-Lekarze Spolka Partnerska, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Med Gastr Sp.z.o.o Sp.k, Lodz
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Centrum Innowacyjnych Terapii, Piaseczno
  - Clinical Research Center Spółka z Ograniczoną Odpowiedzialnością, Medic-R Spółka Komandytowa, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Sonomed Sp. z o.o., Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość
  - Szpital Specjalistyczny sw Lukasza - Oddzial Gastroenterologii, Gmina Końskie, Świętokrzyskie Voivodeship
- Romania (11):
  - Cluj-Napoca Emergency Clinical County Hospital, Cluj-Napoca, Cluj
  - Dr.Carol Davila Emergency University Central Military Hospital, Bucharest
  - Sana Monitoring SRL, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Centrul Medical Hifu Terramed Conformal S.R.L., Bucharest
  - Affidea Romania SRL, Constanța
  - Gastromedica SRL, Iași
  - Dr. Tirnaveanu Amelita Private Practice, Oradea
  - Dr. Goldis Gastroenterology Center SRL, Timișoara
- Russia (17):
  - Kazan State Medical University, Kazan'
  - Moscow Clinical Scientific Center, Moscow
  - Moscow Regional Research Clinical Institute Na Mfvladimirskiy, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Research Institute of Physiology and Basic Medicine, Novosibirsk
  - Rostov State Medical University, Rostov-on-Don
  - Union Clinic, LLC, Saint Petersburg
  - St. Elizabeth Municipal Clinical Hospital, Saint Petersburg
  - First St. Petersburg State Medical University n.a. I.P Pavlov, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Medical University Reaviz, Samara
  - Private Healthcare Institution Clinical Hospital RZD-Medicina of Samara city, Samara
  - Medical Company Hepatolog, LLC, Samara
  - SHI Regional Clinical Hospital, Saratov
  - Smolensk Regional Clinical Hospital, Smoensk
  - Stavropol State Medical University, Stavropol
  - Regional Consulting and Diagnostics Centre, Tyumen
- Serbia (4):
  - Clinical Hospital Center ''Bezanijska Kosa'', Belgrade
  - University Clinical Center Nis, Niš
  - General Hospital Vrsac, Vršac
  - University Clinical Center Kragujevac, Kragujevac, Šumadijski Okrug
- South Africa (3):
  - CLINRESCO, ARWYP Medical Suites, Johannesburg, Gauteng
  - Dr. J Breedt, Pretoria, Gauteng
  - Dr JP Wright, Claremont, Western Cape
- United Kingdom (9):
  - Fairfield General Hospital - PPDS, Lancashire, Bury
  - Pennine Acute Hospitals Trust, Lancashire, Bury
  - Whipps Cross University Hospital, London, London, City of
  - North Tyneside General Hospital, North Shields, Northumberland
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - Aberdeen Royal Infirmary - PPDS, Aberdeen
  - Western General Hospital Edinburgh - PPDS, Edinburh
  - Royal Gwent Hospital - PPDS, Newport
  - New Cross Hospital, Wolverhampton

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fdc4db2bf003ab4733d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 192 sites between 9 February 2018 (first participant first visit) and 23 October 2020 (last participant last visit).
Pre-assignment Details: A total of 380 subjects were enrolled and randomized, of which 378 subjects received the study treatment in this study.
Groups:
- Placebo: Participants received placebo matched to ontamalimab (SHP647) subcutaneous (SC) injection, using a prefilled syringe (PFS) on Week 0, Week 4, and Week 8 in a 12-week treatment period.
- Ontamalimab 25 mg: Participants received 25 milligrams (mg) of ontamalimab (SHP647) SC injection, using a PFS on Week 0, Week 4 and Week 8 in a 12-week treatment period.
- Ontamalimab 75 mg: Participants received 75 mg of ontamalimab (SHP647) SC injection, using a PFS on Week 0, Week 4 and Week 8 in a 12-week treatment period.
Period: Overall Study
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Started | 76 | 153 | 151
Treated | 76 | 151 | 151
Completed | 66 | 136 | 138
Not Completed | 10 | 17 | 13
Not completed — Adverse Event | 3 | 8 | 5
Not completed — Withdrawal by Subject | 4 | 2 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Deviation | 0 | 3 | 2
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Randomized but never treated | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all participants who had received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg | Total
Number analyzed (Participants) | 76 | 151 | 151 | 378
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (13.33) | 39.4 (13.90) | 41.2 (14.75) | 39.9 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 56 | 62 | 151
  Male | 43 | 95 | 89 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 74 | 149 | 146 | 369
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian: Japanese | 1 | 6 | 8 | 15
  Race: Asian: Korean | 0 | 0 | 0 | 0
  Race: Asian: Other | 0 | 4 | 1 | 5
  Race: Black or African American | 1 | 2 | 5 | 8
  Race: White | 72 | 134 | 136 | 342
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Multiple | 2 | 4 | 1 | 7
  Race: Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Remission at Week 12
Description: Remission was defined as a composite score of patient-reported symptoms using daily e-diary and centrally read endoscopy as stool frequency sub-score of 0 or 1 with at least a 1-point change from baseline, rectal bleeding sub-score of 0 and endoscopic sub-score of 0 or 1 (modified, excluded friability). The composite score was a recommended measure consisted of the Mayo score without the physician global assessment (PGA) sub-score and ranged from 0 to 9 points. The Mayo score was a measure of Ulcerative Colitis (UC) disease activity. It ranged from 0 to 12 points and consisted of 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease. The sub-scores were stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: Full analysis set (FAS) consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 12 | 28 | 45
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.617, Cochran-Mantel-Haenszel; P-value was based on Cochran-Mantel-Haenszel chi-square test stratified by actual status of prior anti-TNF treatment and glucocorticoid at baseline
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.018, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission was defined by centrally read endoscopic sub-score 0 or 1 (modified, excluded friability). The centrally read endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 16 | 42 | 62
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.253, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Clinical Remission at Week 12
Description: Clinical remission was defined by stool frequency (SF) sub-score of 0 or 1 with at least a 1-point change from baseline in stool frequency sub-score, and rectal bleeding sub-score of 0. Rectal bleeding is assessed on a scale from 0-3, where 0: no blood seen, 1: streaks of blood with stool less than half time, 2: obvious blood or streaks of blood with stool most of the time, and 3: blood alone passes. Stool frequency is assessed on a scale from 0-3, where 0: normal number of stools for this participant, 1: 1 to 2 stools more than normal, 2: 3 to 4 stools more than normal, and 3: 5 or more stools more than normal. Higher scores indicated more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 29 | 61 | 76
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.764, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.080, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Clinical Response Based on Composite Score at Week 12
Description: Clinical response based on composite score was defined as a decrease from baseline in the composite score of patient-reported symptoms using daily e-diary and centrally read endoscopy of at least 2 points and at least 30 percent (%), with an accompanying decrease in the sub-score for rectal bleeding greater than or equal to (>=) 1 point or a sub-score for rectal bleeding less than or equal to (<=) 1. The composite score was a recommended measure derived from the Mayo score without the PGA sub-score and ranged from 0 to 9 points. The Mayo score was a measure of UC disease activity. It ranged from 0 to 12 points and consisted of 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease The sub-scores were stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 34 | 76 | 99
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.440, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Mucosal Healing Based on Endoscopic and Histological Assessment Using the Geboes Score Grading System at Week 12
Description: Mucosal healing was defined by centrally read endoscopic sub-score 0 or 1 (modified, excluded friability) and centrally read Geboes score of <=2. The centrally read endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease. Geboes score grading system was a validated score for evaluating histologic disease activity in UC as follows: Grade 0 equal to (=) structural and architectural changes; Grade 1 = chronic inflammatory infiltrate; Grade 2 = lamina propria neutrophils and eosinophils; Grade 3 = neutrophils in the epithelium; Grade 4 = crypt destruction; Grade 5 = erosions or ulceration. A higher Geboes score indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 13 | 35 | 51
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.286, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Remission Based on Total Mayo Score at Week 12
Description: Remission was defined as a total Mayo score of <=2 with no individual sub-score (stool frequency, rectal bleeding, endoscopy [modified, excluded friability], and PGA) exceeding 1. The Total Mayo score ranged from 0 to 12 points and consisted of 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 11 | 25 | 40

7. Secondary Outcome: Number of Participants With Clinical Response Based on Total Mayo Score at Week 12
Description: Clinical response (Mayo) was defined as a decrease from baseline in the total Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the sub-score for rectal bleeding >=1 point or an absolute sub-score for rectal bleeding <=1. The Total Mayo score ranged from 0 to 12 points and consisted of the following 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 32 | 78 | 97

8. Secondary Outcome: Number of Participants With Partial Mayo Score <=2 With no Individual Sub-score Greater Than (>) 1 at Weeks 4, 8, and 12
Description: The partial Mayo score ranged from 0 to 9 points and consisted of the following 3 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: Stool frequency (0-3); Rectal bleeding (0-3); PGA (0-3). The partial Mayo score did not include the endoscopy sub-score.
Time Frame: At Weeks 4, 8, and 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants
  At Week 4 | 13 | 38 | 47
  At Week 8 | 23 | 57 | 62
  At Week 12 | 22 | 60 | 78

9. Secondary Outcome: Number of Participants With Clinical Remission With Stool Frequency Sub-scores of 0 or 1 and Rectal Bleeding Sub-score of 0 at Weeks 4 and 8
Description: Clinical remission was defined as stool frequency sub-score of 0 or 1 with at least a 1-point change from baseline in stool frequency sub-score, and a rectal bleeding sub-score of 0. Rectal bleeding was assessed on a scale from 0-3, where 0: no blood seen, 1: streaks of blood with stool less than half time, 2: obvious blood or streaks of blood with stool most of the time, and 3: blood alone passes. Stool frequency was assessed on a scale from 0-3, where 0: normal number of stools for this participant, 1: 1 to 2 stools more than normal, 2: 3 to 4 stools more than normal, and 3: 5 or more stools more than normal. Higher scores indicated more severe disease
Time Frame: At Weeks 4 and 8
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants
  At Week 4 | 15 | 34 | 38
  At Week 8 | 23 | 57 | 60

10. Secondary Outcome: Number of Participants With Endoscopic Remission With Sub-score of 0 at Week 12
Description: Endoscopic remission was defined by centrally read endoscopic sub-score 0 (modified, excluded friability). The centrally read endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 9 | 10 | 22

11. Secondary Outcome: Number of Participants With Clinical Remission With Both Rectal Bleeding and Stool Frequency Sub-scores of 0 at Weeks 4, 8, and 12
Description: Clinical remission was defined as both rectal bleeding and stool frequency sub-scores of 0. Rectal bleeding was assessed on a scale from 0-3, where 0: no blood seen, 1: streaks of blood with stool less than half time, 2: obvious blood or streaks of blood with stool most of the time, and 3: blood alone passes. Stool frequency was assessed on a scale from 0-3, where 0: normal number of stools for this participant, 1: 1 to 2 stools more than normal, 2: 3 to 4 stools more than normal, and 3: 5 or more stools more than normal. Higher scores indicated more severe disease.
Time Frame: At Weeks 4, 8, and 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants
  At Week 4 | 7 | 20 | 15
  At Week 8 | 12 | 24 | 29
  At Week 12 | 11 | 37 | 39

12. Secondary Outcome: Number of Participants With Deep Remission at Week 12
Description: Deep remission was defined as both endoscopic and rectal bleeding sub-scores of 0, and stool frequency sub-score <=1 and a centrally read Geboes score of <=2. The stool frequency sub-score, rectal bleeding sub-score and endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease. The composite score was a recommended measure consisted of the Mayo score without the PGA sub-score and ranged from 0 to 9 points. Geboes score grading system was a validated score for evaluating histologic disease activity in UC as follows: Grade 0 = structural and architectural changes; Grade 1 = chronic inflammatory infiltrate; Grade 2 = lamina propria neutrophils and eosinophils; Grade 3 = neutrophils in the epithelium; Grade 4 = crypt destruction; Grade 5 = erosions or ulceration. A higher Geboes score indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants | 7 | 6 | 18

13. Secondary Outcome: Change From Baseline in Average Worst Abdominal Pain Score Based on Patient Reported Outcome-ulcerative Colitis (PRO-UC) Daily e-Diary at Week 12
Description: PRO-UC daily e-diary data was collected using a daily e-diary during the treatment period. Collection of the daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data of abdominal pain worst severity, as experienced over the previous 24 hours, in the e-diary. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or non-consecutive) of the last 10 days prior to scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Abdominal pain's worst severity assessment was based on an 11-point numerical rating scale with 0 anchor at "No pain" and 10 at "Worst Imaginable Pain" as experienced over the previous 24 hours, in e-diary. Higher scores indicating more severe pain.
Time Frame: Baseline, Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 68 | 136 | 141
Score on a Scale | -1.69 (0.271) | -2.15 (0.196) | -2.14 (0.194)

14. Secondary Outcome: Change From Baseline in Diarrhea (Average Loose Bowel Movements) Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC daily e-diary data was collected using a daily e-diary during the treatment period. Collection of the daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for number of loose bowel movement, as experienced over the previous 24 hours, in the e-diary. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number of loose bowel movement ranged from 0-27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 68 | 136 | 141
Score on a Scale | -2.90 (0.378) | -3.08 (0.273) | -3.50 (0.272)

15. Secondary Outcome: Change From Baseline in Average Bowel Movements With Urgency Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC daily e-diary data was collected using a daily e-diary during the treatment period. Collection of the daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for number of bowel movement with urgency, as experienced over the previous 24 hours. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number bowel movements urgency ranged from 0 to 27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 68 | 136 | 141
Score on a Scale | -2.38 (0.341) | -2.60 (0.246) | -2.84 (0.245)

16. Secondary Outcome: Change From Baseline in Absolute Stool Frequency (Average Number of Bowel Movements) Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC daily e-diary data was collected using a daily e-diary during the treatment period. Collection of the daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for average number of bowel movements, as experienced over the previous 24 hours. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number bowel movements ranged from 0 to 27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 68 | 136 | 141
Score on a Scale | -2.27 (0.363) | -2.78 (0.262) | -2.86 (0.260)

17. Secondary Outcome: Change From Baseline in Absolute Rectal Bleeding (Average Number Bowel Movements With Blood) Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC daily e-diary data was collected using a daily e-diary during the treatment period. Collection of the daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for average number of bowel movements with blood, as experienced over the previous 24 hours. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number bowel movements with blood ranged from 0 to 27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 68 | 136 | 141
Score on a Scale | -2.85 (0.337) | -3.50 (0.242) | -3.50 (0.240)

18. Secondary Outcome: Change From Baseline in Total Sign/Symptom Score Based on PRO-UC Daily e-Diary at Week 12
Description: Total sign/symptom score was the average of the average scores of worst abdominal pain over the past 24 hours and the conversion scale values for number of bowel movements blood, number of bowel movements with urgency, number of bowel movements and number of loose bowel movements, with scale ranged of 0-10, with higher scores indicating higher severity.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 68 | 136 | 141
Score on a Scale | -1.92 (0.234) | -2.15 (0.169) | 0.169 (0.168)

19. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Domains Scores at Weeks 8 and 12
Description: IBDQ was a psychometrically validated participant-reported outcome (PRO) instrument for measuring the disease-specific health-related quality of life (HRQL) in participants with inflammatory bowel disease, including UC. The IBDQ consisted of 32 items, which were grouped into 4 domains: bowel function, emotional status, systemic symptoms, and social function The 4 domains were scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35; Emotional function: 12 to 84; Social function: 5 to 35. Higher scores indicating a better quality of life.
Time Frame: Baseline, Weeks 8 and 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed refer to participants evaluable at given categories.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 72 | 147 | 144
Score on a Scale
  IBDQ Bowel Function Dimension Score: Change at Week 8 | 11.32 (1.414) | 16.27 (1.006) | 15.70 (1.026)
  IBDQ Bowel Function Dimension Score: Change at Week 12: number analyzed (Participants) | 69 | 141 | 142
  IBDQ Bowel Function Dimension Score: Change at Week 12 | 12.89 (1.568) | 16.19 (1.114) | 17.18 (1.127)
  IBDQ Emotional Status Dimension Score: Change at Week 8 | 9.15 (1.596) | 14.54 (1.136) | 14.46 (1.157)
  IBDQ Emotional Status Dimension Score: Change at Week 12: number analyzed (Participants) | 69 | 141 | 142
  IBDQ Emotional Status Dimension Score: Change at Week 12 | 10.10 (1.732) | 14.62 (1.230) | 16.01 (1.243)
  IBDQ Systemic Symptoms Dimension Score: Change at Week 8 | 4.05 (0.681) | 6.47 (0.485) | 6.03 (0.494)
  IBDQ Systemic Symptoms Dimension Score: Change at Week 12: number analyzed (Participants) | 69 | 141 | 142
  IBDQ Systemic Symptoms Dimension Score: Change at Week 12 | 4.44 (0.735) | 6.19 (0.522) | 6.72 (0.528)
  IBDQ Social Function Dimension Score: Change at Week 8 | 4.89 (0.806) | 7.59 (0.576) | 7.14 (0.586)
  IBDQ Social Function Dimension Score: Change at Week 12: number analyzed (Participants) | 69 | 141 | 142
  IBDQ Social Function Dimension Score: Change at Week 12 | 6.11 (0.862) | 7.95 (0.615) | 8.24 (0.621)

20. Secondary Outcome: Change From Baseline in IBDQ Total Scores at Weeks 8 and 12
Description: IBDQ was a psychometrically validated PRO instrument for measuring the disease-specific HRQL in participants with inflammatory bowel disease, included UC. The IBDQ consisted of 32 items, which were grouped into 4 domains: bowel function, emotional status, systemic symptoms, and social function. The 4 domains were scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35; Emotional function: 12 to 84; Social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicating better HRQL. A score of at least 170 corresponds to clinical remission and an increase of at least 16 points was considered to indicate a clinically meaningful improvement.
Time Frame: Baseline, Weeks 8 and 12
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 72 | 147 | 144
Score on a Scale
  Change at Week 8 | 29.55 (4.205) | 44.97 (2.999) | 43.36 (3.053)
  Change at Week 12: number analyzed (Participants) | 69 | 141 | 142
  Change at Week 12 | 33.52 (4.595) | 45.00 (3.269) | 48.12 (3.305)

21. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36), Version 2, Acute (Physical and Mental Component Summary Scores) at Week 12
Description: SF-36 was a generic quality-of-life instrument that had been widely used to assess health-related quality of life (HRQL) of participants). SF-36 consisted of 36 items that were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]). Four domains comprised physical component summary (PCS) score (physical functioning, role-physical, bodily pain, general health) and remaining 4 domains comprised mental component summary (MCS) score (vitality, social functioning, role-emotional, mental health). The scores ranged from 0 to 100. Higher scores indicating better HRQL.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 69 | 141 | 142
Score on a Scale
  Physical Component Summary: Change at Week 12 | 4.92 (0.848) | 6.76 (0.604) | 6.54 (0.610)
  Mental Component Summary: Change at Week 12 | 3.89 (1.113) | 5.83 (0.792) | 6.37 (0.799)

22. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36), Version 2, Acute (Individual Domain Scores) at Week 12
Description: SF-36 was a generic quality-of-life instrument that had been widely used to assess HRQL of participants. The SF-36 consisted of 36 items that were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]), with scores ranged from 0 to 100. Higher scores indicating better HRQL.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 69 | 141 | 142
Score on a Scale
  Physical Functioning: Change at Week 12 | 4.89 (0.766) | 5.41 (0.545) | 4.32 (0.550)
  Role-Physical: Change at Week 12 | 3.99 (1.059) | 6.97 (0.754) | 7.65 (0.762)
  Bodily Pain: Change at Week 12 | 6.28 (1.132) | 8.83 (0.805) | 8.50 (0.814)
  General Health: Change at Week 12 | 3.36 (0.976) | 4.78 (0.693) | 5.36 (0.699)
  Vitality: Change at Week 12 | 4.96 (1.202) | 8.08 (0.857) | 8.69 (0.865)
  Social Functioning: Change at Week 12 | 6.07 (1.160) | 7.80 (0.827) | 8.56 (0.833)
  Role-Emotional: Change at Week 12 | 3.25 (1.082) | 4.55 (0.765) | 4.04 (0.772)
  Mental Health: Change at Week 12 | 3.93 (1.096) | 5.81 (0.781) | 6.59 (0.786)

23. Secondary Outcome: Number of Participants Based on In-patient Hospitalization
Description: Number of participants based on inpatient hospitalization due to all-cause hospitalization, gastrointestinal related, other illness/problem, and who had undergone gastrointestinal related procedures during the entire study period was reported.
Time Frame: Baseline up to Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 76 | 151 | 151
Participants
  All-Cause Hospitalization | 3 | 8 | 5
  Gastrointestinal Related | 0 | 5 | 2
  Other Illness/Problem | 3 | 3 | 3
  Undergo Gastrointestinal Related Procedures | 0 | 5 | 2

24. Secondary Outcome: Median Duration of Total In-patient Days
Description: In-patient days were calculated as Date of discharge - Date of admission + 1. Median duration of total inpatient days during the entire study period was reported.
Time Frame: Baseline up to Week 12
Population: as for outcome 13
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 3 | 8 | 5
Days | 5.0 [3 to 7] | 7.0 [1 to 13] | 4.0 [3 to 8]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Week 29)
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/151 | 1/151
Serious Adverse Events (participants affected / at risk) | 5/76 | 10/151 | 8/151
Other Adverse Events (participants affected / at risk) | 10/76 | 20/151 | 6/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Ontamalimab 25 mg (N=151) | Ontamalimab 75 mg (N=151)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Ontamalimab 25 mg (N=151) | Ontamalimab 75 mg (N=151)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 10 (11) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 10 (10) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated early as per the sponsor decision to discontinue the ontamalimab clinical trial development program for inflammatory bowel diseases (IBD) for reasons unrelated to safety and efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT03259334/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03259334/SAP_001.pdf